CLINICAL TRIAL: NCT05344729
Title: A Randomized, Open-label, Single-center, Two-period, Two-crossover Phase I Clinical Trial to Evaluate the Effect of Food on the Pharmacokinetics of TQB3616 Capsules in Healthy Adult Subjects
Brief Title: Clinical Trial for Effect of TQB3616 Capsule on Pharmacokinetics in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TQB3616-I-02
Record Dates: First submitted 2022-04-01; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Recurrent/Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB3616 Capsule- Fasted+ TQB3616 Capsule- After meal (Experimental): Subjects in Arm A will take TQB3616 capsules under fasting and fed state in Cycle 1 and Cycle 2, respectively
  Interventions: Drug: TQB3616 Capsule
- TQB3616 Capsule- After meal + TQB3616 Capsule- Fasted (Experimental): Subjects in Arm B will take TQB3616 capsules in Cycle 1 and Cycle 2 under fasting state, respectively
  Interventions: Drug: TQB3616 Capsule

INTERVENTIONS:
Drug: TQB3616 Capsule — It inhibits the proliferation of tumor cells by reducing the level of retinoblastoma protein (Rb) phosphorylation in cancer cells and blocking the progression of cells from G1 to S phase.

SUMMARY:
TQB3616 capsule is a small molecule oral drug developed by Chia Tai Tianqing Pharmaceutical Group Co., Ltd., which inhibits cyclin-dependent kinases 4 and 6 (CDK4/6). Its main mechanism of action is to inhibit the proliferation of tumor cells by reducing the phosphorylation level of retinoblastoma protein (Rb) in cancer cells and blocking the progression of cells from G1 phase to S phase. This study is a randomized, open-label, single-center, two-period, two-crossover phase I clinical trial to assess the effect of food on the pharmacokinetics of TQB3616 capsules in healthy adult subjects, to evaluate the effect of food on the pharmacokinetics of TQB3616 capsules after oral administration in healthy adult Chinese subjects and to observe the safety of TQB3616 capsules after single oral administration in healthy subjects.Each subject will be randomly assigned to one of two groups (group A and B). A total of 16 subjects were enrolled, all taking TQB3616 capsules 180mg, including 8 subjects in group A and 8 subjects in group B. The study included screening period, randomization, first cycle, washout period and second cycle. The first cycle and second cycle each contained 3 return visits. 18 pharmacokinetic samples were collected every cycle for pharmacokinetic index analysis. Vital signs, physical examinations, 12-lead electrocardiograms, clinical laboratory tests, adverse events, drug combination and non-drug therapy information were collected during the study to ensure the safety of the subjects.

ELIGIBILITY:
Inclusion Criteria:

* 1 Sign the informed consent form before the trial and fully understand the content, process and possible adverse reactions of the trial;
* 2 Be able to complete the study according to the requirements of the study protocol;
* 3 Subjects aged 18 to 65 years (including 18 and 65 years);
* 4 Body mass index (BMI) ≥ 18 and ≤ 28 kg/m2, and male body weight ≥ 50 kg Female body weight ≥ 45 kg;
* 5 Health condition: no mental disorders, no history of cardiovascular system, nervous system, respiratory system, digestive system, urinary system, endocrine system and metabolic abnormalities;
* 6 Subjets had no plans to become pregnant and voluntarily took effective contraceptive measures from 2 weeks before dosing to at least 6 months after the last dose of study drug.

Exclusion Criteria:

* 1 Patients with a history of neuropsychiatric, respiratory, cardiovascular, gastrointestinal, hemolymphatic, hepatic or renal insufficiency, endocrine, musculoskeletal system disease or other diseases, which may affect drug metabolism or safety as judged by the investigator;
* 2 Allergic constitution or previous history of two or more kinds of food or drug allergy;
* 3 Hyperactive/venous thrombotic events within 6 months, such as cerebrovascular accident (including temporary ischemic attack), deep venous thrombosis and pulmonary embolism;
* 4 Patients with multiple factors affecting oral drugs (such as inability to swallow, gastrointestinal diseases);
* 5 Taking any prescription drugs, over-the-counter drugs, vitamin products or herbal medicines within 1 month before taking the study drug;
* 6 Administration of CYP3A4 inhibitors or inducers within 1 month before screening or before study drug;
* 7 Taking special diet (including grapefruit, etc.) or strenuous exercise, or other factors affecting drug absorption, distribution, metabolism, excretion, etc. within 14 days before screening;
* 8 Abnormal and clinically significant laboratory findings during the screening period;
* 9 Blood donation or significant blood loss (> 450 mL) within 3 months prior to administration of study drug;
* 10 Participated in any drug clinical trial within 3 months before taking the study drug;
* 11 Smoking more than 5 cigarettes per day within 3 months before the trial;
* 12 Positive breath alcohol test or history of alcoholism (14 units of alcohol per week: 1 unit = 360 mL of beer or 45 mL of spirits with 40% alcohol or 150 mL of wine);
* 13 Drug screening positive or drug use 3 months before the trial;
* 14 Inability to tolerate venipuncture for blood sampling or poor vascular status;
* 15 Subjets cannot complete the trial due to personal reasons;
* 16 Other conditions considered inappropriate by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Peak concentration(Cmax) | The first and second cycles before administration, 1, 2, 3, 4, 5, 5.5, 6, 6.5, 7, 8, 12, 24, 48, 72, 120, 168 and 264 hours after administration (each cycle is 12 days)
  Maximum plasma drug concentration
Area under the time-concentration curve from 0 to t hours after drug administration(AUC0-t)) | The first and second cycles before administration, 1, 2, 3, 4, 5, 5.5, 6, 6.5, 7, 8, 12, 24, 48, 72, 120, 168 and 264 hours after administration (each cycle is 12 days)
  Area under the plasma concentration-time curve from the time of first dose to the time of the last measurable concentration
Area under the time-concentration curve from 0 to infinity after drug administration(AUC0-∞) | The first and second cycles before administration, 1, 2, 3, 4, 5, 5.5, 6, 6.5, 7, 8, 12, 24, 48, 72, 120, 168 and 264 hours after administration (each cycle is 12 days)
  Area under the plasma concentration-time curve from the time of first dosing extrapolated to infinity

SECONDARY OUTCOMES:
Time to peak(Tmax) | The first and second cycles before administration, 1, 2, 3, 4, 5, 5.5, 6, 6.5, 7, 8, 12, 24, 48, 72, 120, 168 and 264 hours after administration (each cycle is 12 days)
  Time to reach maximum (peak) plasma concentration following drug administration
Elimination half-life(t1/2) | The first and second cycles before administration, 1, 2, 3, 4, 5, 5.5, 6, 6.5, 7, 8, 12, 24, 48, 72, 120, 168 and 264 hours after administration (each cycle is 12 days)
  Elimination half-life (to be used in one-or non-compartmental model)
Apparent volume of distribution(Vd/F) | The first and second cycles before administration, 1, 2, 3, 4, 5, 5.5, 6, 6.5, 7, 8, 12, 24, 48, 72, 120, 168 and 264 hours after administration (each cycle is 12 days)
  Apparent volume of distribution after non-intravenous administration
Apparent clearance(CL/F) | The first and second cycles before administration, 1, 2, 3, 4, 5, 5.5, 6, 6.5, 7, 8, 12, 24, 48, 72, 120, 168 and 264 hours after administration (each cycle is 12 days)
  Apparent total clearance of the drug from plasma after oral administration
Bioavailability(F) | The first and second cycles before administration, 1, 2, 3, 4, 5, 5.5, 6, 6.5, 7, 8, 12, 24, 48, 72, 120, 168 and 264 hours after administration (each cycle is 12 days)
  Bioavailability (systemic availability of the administered dose)
Elimination rate constant (λz) | The first and second cycles before administration, 1, 2, 3, 4, 5, 5.5, 6, 6.5, 7, 8, 12, 24, 48, 72, 120, 168 and 264 hours after administration (each cycle is 12 days)
  Terminal disposition rate constant/terminal rate constant
Body temperature | The first and second cycles before adminisyration, 1, 2, 6, 8, 24, 48, 72, 120, 168 and 264 hours after administration (each cycle is 12 days)
  Abnormal body temperature
Pulse | The first and second cycles before adminisyration, 1, 2, 6, 8, 24, 48, 72, 120, 168 and 264 hours after administration (each cycle is 12 days)
  Abnormal pulse
Blood pressure | The first and second cycles before adminisyration, 1, 2, 6, 8, 24, 48, 72, 120, 168 and 264 hours after administration (each cycle is 12 days)
  Abnormal blood pressure
Physical examination | After the end of the first cycle and the second cycle (each cycle is 12 days)
  The doctor percusses, looks, and questions the subject
Electrocardiogram QT interval | After the end of the first cycle and the second cycle (each cycle is 12 days)
  Safety Checks
Adverse Events | Up to 31 days (each cycle is 12 days)
  Monitor the safety indicators of subjects during the trial

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Changchun University of Traditional Chinese Medicine, Changchun, Jilin, China

REFERENCES:
- [Derived] Dai J, Zhou Y, Zhang L, Ren Q, Liu Z, Wang Y, Cheng Y, Deng Q, Yang H, Zhang H. The food effect on the pharmacokinetics of TQB3616 capsule in Chinse healthy subjects: a randomized, open-label, single-center, two-period, two-sequence crossover phase I clinical trial. Front Pharmacol. 2025 May 30;16:1586368. doi: 10.3389/fphar.2025.1586368. eCollection 2025. PMID 40520159